CLINICAL TRIAL: NCT04241887
Title: Is Thoracic Paravertebral Block a Better Option Than Conscious Sedation for Percutaneous Radiofrequency Ablation of Liver Tumors
Brief Title: Is Thoracic Paravertebral Block a Better Option Than Conscious Sedation for PRFA of Liver Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warmia and Mazury (Other)
Responsible Party: Principal Investigator, Malgorzata Braczkowska, Principal Investigator, University of Warmia and Mazury
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UWarmiaMazury-2
Record Dates: First submitted 2020-01-17; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Liver Tumor
Keywords: Paravertebral block; Anaesthesia; Analgesia; regional anaesthesia; pain; patient satisfaction; patient comfort; operator satisfaction
MeSH Terms: conditions — Carcinoma, Hepatocellular; Agnosia; Pain; Patient Satisfaction | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: 30 patients scheduled for an elective Percutaneus Radiofrequency Ablation (PRFA) of a hepatocellular carcinoma were enrolled in the study. Patients were divided in 2 groups:
  * group PVB - 15 patients under paravertebral block anaesthesia
  * group BB - 15 patients under local anesthesia, without paravertebral block.
Who Masked: Participant
Masking Description: Participants were randomly assigned into 2 groups (computerized randomization program).
  group PVB - patients under paravertebral block anesthesia, group BB - patients under local anesthesia, without paravertebral block.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group PVB (Experimental): standard analgosedation + paravertebral thoracic blockade with 20 ml 0.25% bupivacaine (Bupivacainum hydrochloricum WZF 0,5%, Polfa warszawa S.A.)
  Interventions: Procedure: thoracic paravertebral blockade
- group BB (Active Comparator): standard analgosedation + local anesthesia of the skin and subcutaneous tissue with 5ml 0,5% lignocaine (Lignocainum hydrochlorici, WZF 1%).
  Interventions: Procedure: local anaesthesia

INTERVENTIONS:
Procedure: thoracic paravertebral blockade — Anesthesia was performed under the ultrasound guidance: the Th8 spinous process was identified, then a probe was moved lateral to medial until two adjacent transverse processes and the pleura were visible. After anaesthetising the skin with 2ml of 1% lignocaine (Lignocainum hydrochlorici, WZF 1%), the Touhy needle 22G (Smith Medical)was introduced under the real time guidance. Once in the paravertebral space, 20ml of 0,25% bupivacaine (Bupivacainum hydrochloricum WZF 0,5%, Polfa Warsaw SA) was injected with an end point of a characteristic pleural displacement.
  Arms: group PVB
Procedure: local anaesthesia — Local infiltration anaesthesia with 0.5% lignocaine 5ml (Lignocainum hydrochlorici, WZF 1%) was applied to the skin and the potential needle path of ablation.
  Arms: group BB

SUMMARY:
Percutaneus radiofrequency ablation (RFA) of liver tumors causes acute pain during the periooperative setting. In order to facilitate tumor access, patient should collaborate with a surgeon during the procedurę, therefore should be conscious.

This study aims to assess the impact of a single shot thoracic paravertebral block (TPVB) on a patient's haemodynamic stability, patient's and operator's comfort and satisfaction during the operation and analgesia in the post-operative period.

DETAILED DESCRIPTION:
High temperatures used during the percutaneus radiofrequency ablation (PRFA) of liver tumors can cause acute pain in the perioperative setting. In order to facilitate tumor exposure and access, patient should collaborate with a surgeon during the procedurę, therefore should be conscious. It is mandatory to provide an adequate acute postoperative pain control for our patients.

This prospective randomized, single center study was approved by the Bioethics Committee at the University of Warmia and Mazury in Olsztyn, (Poland) under the resolution No. 46/2017.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary liver tumor (HCC)
* patient scheduled for an elective surgery
* tumor diameter) <5 cm two tumors <3cm
* Age >18 years
* Physical State 1,2 or 3 of the American Society of Anesthesiology (ASA)

Exclusion Criteria:

* ASA IV and V
* Thrombocytopenia (<40x10 ^ 9 / L)
* Severe cirrhosis (Child-Pugh C classification)
* History of psychiatric/cognitive disease
* Patients who do not give informed consent
* Patients with contraindications or history of hypersensitivity to local anaesthesia drugs
* History of chronic pain, chronic opioid use (> 3 months)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of PVB on pain intensity | NRS during the procedure and 0,1,3,6,24 hours post surgery
  The level of pain will be assessed in all groups (PVB and BB) basing on the NRS scale (NRS 0- no pain, NRS 10 - the worst pain imaginable) Self reported pain intensity in 5 time points based on the numerical rating scale NRS (where 0 is no pain, 10 is the strongest pain).
  comparison of analgesic drug use in both groups
Effectiveness of PVB on pain intensity | 0,1,3,6,24 hours post surgery
  The level of pain will be assessed in all groups (PVB and BB) basing on analgesic drugs consumption

SECONDARY OUTCOMES:
Patients' satisfaction | 24 hours post surgery
  Patients' satisfaction will be assessed in all groups (PVB and BB) basing on a survey
Surgeon's satisfaction | 0 h post surgery (immediately after surgery)
  Surgeon's satisfaction will be assessed in all groups (PVB and BB) basing on a survey (where 0 is no satisfaction, 10-maximal satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Mayzner-Zawadzka, PhD, Study Chair — University of Warmia and Mazury Faculty of Medicine (University Hospital)
Locations (1):
- Anesthesiology and Intensive Care Clinical Ward, Clinical University Hospital, Olsztyn, Warmian-Masurian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified study participants data for all primary and secondary outcome measures
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 12 months of study completion
Access Criteria: Data will be made available for researchers who provide a methodologically sound proposal. Proposals should be directed to m.braczkowska@gmail.com . Data access requests will be reviewed by an External Independent Review Panel. To gain access, data requestors will need to sign a data access agreement.